CLINICAL TRIAL: NCT06608394
Title: Effect of Preoperative Exercise Habits on Knee Function and Recurrence Rate After Anterior Cruciate Ligament Reconstruction
Status: Recruiting | Type: Observational
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: M2024765
Record Dates: First submitted 2024-09-19; First posted 2024-09-23 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2024-09

CONDITIONS: Anterior Cruciate Ligament Rupture
Keywords: anterior cruciate ligament injuries; exercise habit
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (4):
- Preoperative exercise habits group: Moderate-intensity aerobic exercise or strength training was performed at least 3 times per week for 6 months before surgery.
  Interventions: Other: no intervention
- No exercise habit before operation group: There was no regular exercise habit for 6 months before surgery
  Interventions: Other: no intervention
- The exercise habit group was maintained after operation: Moderate-intensity aerobic exercise was continued at least three times per week after surgery
  Interventions: Other: no intervention
- The exercise habit was not maintained after operation: Did not maintain a regular exercise habit after surgery
  Interventions: Other: no intervention

INTERVENTIONS:
Other: no intervention — no intervention

SUMMARY:
The aim of this study is to compare the knee function between patients with and without preoperative exercise habits at 1, 2 and 5 years after ACL surgery, and further analyze the effect of maintaining exercise habits on knee function and recurrence rate

DETAILED DESCRIPTION:
Objective:

1. To compare the knee function between active and inactive patients at 1, 2, and 5 years after ACL surgery.
2. To investigate the difference of knee function and recurrence rate between patients with and without postoperative exercise habit.

Methods: This is a single-center, controlled follow-up cohort study. Inclusion criteria included patients aged 18-45 years with confirmed ACL injury who were scheduled to undergo ACL reconstruction surgery. Exercise habits were recorded before operation, and knee joint function and exercise level were evaluated by questionnaires. All patients received standardized ACL reconstruction surgery and rehabilitation program after surgery. In prospective cohort study, 121 patients were divided into running group and non-running group according to their preoperative exercise habits. At 3 months after surgery, running was included in the rehabilitation program, and the patients were further divided into postoperative running and non-running groups and followed up for one year.In Postoperative cohort study， follow-up was collected and evaluated at 1 year, 2 years and 5 years, including knee function, exercise level and recurrence. The study was divided into four groups: preoperative running group , preoperative non-running group , preoperative and postoperative running group and preoperative non-running and postoperative running group to analyze the effects of preoperative and postoperative exercise habits on knee joint function and recurrence rate. The results of this study will help to deepen the understanding of the impact of preoperative exercise habits and postoperative exercise maintenance on knee function and recurrence rate after ACL reconstruction, and then provide guidance for clinical practice, optimize postoperative rehabilitation programs, and ultimately improve the quality of life of patients.

Subjects: Patients with anterior cruciate ligament rupture in Department of Sports Medicine, Peking University Third Hospital 1.1.1 Inclusion criteria

1. Age of 18-45 years old, male or female.
2. Patients were diagnosed with anterior cruciate ligament injury and planned to undergo anterior cruciate ligament reconstruction surgery 1.1.2 Exclusion criteria Presence of other severe knee disorders (e.g., arthritis).

   * Prior history of other knee surgeries
   * Inability to complete a postoperative rehabilitation program or long-term follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Patients with anterior cruciate ligament rupture in Department of Sports Medicine, Peking University Third Hospital

Exclusion Criteria:

* Severe other knee disorders (e.g., arthritis) are present.
* Prior history of other knee surgeries
* Inability to complete a postoperative rehabilitation program or long-term follow-up

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: An ACL injury was diagnosed and an ACL reconstruction surgery was planned
Sampling Method: Probability Sample
Enrollment: 361 (Estimated)
Dates: Start 2024-11-30 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Lysholm knee score | 1year，2year，5year
IKDC score | 1year，2year，5year
Tegner score | 1year，2year，5year
Beighton Score | 1year，2year，5year

SECONDARY OUTCOMES:
recurrence rate | 1year，2year，5year

CONTACTS AND LOCATIONS:
Locations (1):
- Peking university third hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No